CLINICAL TRIAL: NCT03454906
Title: Baskent University Nephrology Department
Brief Title: Factors Influencing Hemoglobin Variability and Its Association With Mortality in Hemodialysis Patients
Status: Completed | Type: Observational
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, Zeynep Bal, Baskent University Nephrology Department, Baskent University
Other Study IDs: KA09/358
Record Dates: First submitted 2018-02-02; First posted 2018-03-06 (Actual); Last update posted 2018-03-06 (Actual); Status verified 2018-02

CONDITIONS: Hemodialysis-Induced Symptom
Keywords: hemodialysis; hemoglobin variability; mortality; nutrition; inflammation
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- L Hemoglobin: L Hemoglobin: consistently low all 6 months with low hemoglobin levels
- T Hemoglobin: T Hemoglobin; consistently within the target range all 6 months with target-range hemoglobin levels
- H Hemoglobin: H Hemoglobin: consistently high all 6 months with high hemoglobin levels
- LAL Hemoglobin: LAL Hemoglobin: low amplitude fluctuation with low hemoglobin; all 6 months with low or target range hemoglobin levels
- LAH Hemoglobin: LAH Hemoglobin: low-amplitude fluctuation with high hemoglobin levels 6 months with target-range or high hemoglobin levels)
- HA Hemoglobin: HA Hemoglobin ; high-amplitude fluctuation low, target-range, and high hemoglobin levels within the 6 month period

SUMMARY:
The aim of the study is to investigate the factors influencing hemoglobin variability with inflammatory and nutritional parameters and its associations with all-cause mortality among hemodialysis patients.

DETAILED DESCRIPTION:
Fluctuation in hemoglobin levels that is known as hemoglobin variability during treatment with ESA is a well-documented phenomenon. Several factors have been found to affect hemoglobin variability, including drug related, such as pharmacokinetic parameters, patient-related differences in demographic characteristics and factors affecting clinical status, as well as clinical practice guidelines, treatment protocols and reimbursement policies. Inflammation is also an important factor associated with hemoglobin variability, and the consequences of persistent inflammatory activity are far-reaching in affected patients.

In present study, the factors influencing hemoglobin variability with inflammatory and nutritional parameters and its associations with all-cause mortality among hemodialysis patients are investigated.

ELIGIBILITY:
Inclusion Criteria:

* Age >18
* on chronic hemodialysis treatment

Exclusion Criteria:

* All patients had a minimum of six hemoglobin measurements within a 6- month period, and they were excluded if they received a kidney transplant during this period or those who had blood transfusions during the baseline period.
* Patients with serum ferritin<100 μg/L were also excluded from the study because of reimbursement of our country.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: -one hundred and sixty nine patient that receive chronic hemodialysis treatment in Baskent university hospital were enrolled to the study.
Sampling Method: Non-Probability Sample
Enrollment: 169 (Actual)
Dates: Start 2009-01 (Actual); Primary Completion 2010-01 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Factors Influencing Hemoglobin Variability and Its Association with Mortality in Hemodialysis Patients | six month
  investigation of factors influencing hemoglobin variability with inflammatory and nutritional parameters and the association of hemoglobin variability with all-cause mortality among hemodialysis patients

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bal Z, Demirci BG, Karakose S, Tutal E, Erkmen Uyar M, Acar NO, Sezer S. Factors Influencing Hemoglobin Variability and Its Association with Mortality in Hemodialysis Patients. ScientificWorldJournal. 2018 Apr 1;2018:8065691. doi: 10.1155/2018/8065691. eCollection 2018. PMID 29805324